CLINICAL TRIAL: NCT06027905
Title: Novartis - Closing the Gap in Cardiovascular Risk: Engage, Empower, Evaluate
Acronym: E3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22123002; 1036009 (Other Grant/Funding Number: Novartis Pharmaceuticals)
Record Dates: First submitted 2023-08-21; First posted 2023-09-07 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: hypertension; self-monitoring; social determinants of health; adherence
MeSH Terms: conditions — Hypertension | interventions — Social Work

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Blood Pressure Monitoring and Social Intervention (Experimental): Participants are enrolled in a remote blood pressure monitoring program and social intervention composed of remote outreach from a team of community health worker, pharmacist, nurse, and social worker for 12 weeks.
  Interventions: Other: E3 Remote Monitoring and Social Intervention

INTERVENTIONS:
Other: E3 Remote Monitoring and Social Intervention — Patients are enrolled in a 12 week remote blood pressure monitoring program composed of a community health worker, nurse, pharmacist and social worker. Participants will receive a home cellular blood pressure cuff for remote monitoring and will receive tele-health calls from their community health worker to assist with blood pressure taking technique and adherence, medication adherence, education around diet and activity. Social work is available to provide institutional and community resources to patients with social needs. Patients will be screened pre intervention and post intervention for medication adherence and social determinants of health needs. The team nurse monitors and triages home blood pressures on the remote portal. The pharmacist assists with medication reconciliation, adherence, and titration of medications according to standards or care.

SUMMARY:
This study aims to decrease the racial gap in high blood pressure in African American and Latinx patients in Rush University Medical Center clinics.

DETAILED DESCRIPTION:
The study is a clinic-based study with remote patient monitoring that uses a team based intervention composed of community health worker (CHW), nurse (RN), pharmacist, and social worker (SW). Eligible patients are those who are 18 years old and over, African American and/or LatinX with elevated CVD risk starting with stage II hypertension following with a primary care provider in an eligible Rush primary care clinic who have access to a phone or device with call or video capabilities in their home. Eligible patients will be enrolled in the study by their participating Rush clinician via two methods: 1) encountering eligible patients during a clinic visit and enrolling them directly into the program with a community health worker (CHW); 2) generating a list of eligible elevated CVD risk patients and CHWs remotely calling patients to enroll in the program. Patients enrolled in the program will receive the intervention of additional resources for improvement of cardiovascular risk in addition to usual care.

For patients who are enrolled with a CHW onsite, the patient will proceed directly to a visit with the CHW. During the CHW visit, the patient will be introduced to the program, and will undergo verbal consent for the program. Screening for the social determinants of health (SDOH) (using the clinic questionnaire already in use at all Rush primary care clinics) will be completed if not already completed prior to the clinic visit. If patients screen positive for more than three social determinants of health needs, or if they screen positive for homelessness or violence independently, they will be referred to the program social worker who will proceed with a tailored social work intervention remotely during the 3 month course of the study. Patients will also complete the ARMS (Adherence to Refills and Medications Scale) medication adherence screening questionnaire, and receive a cellular enable blood pressure cuff provided from the company HealthSnap. The CHW will provide training on usage of the cuff and enroll the patient in the remote monitoring HealthSnap dashboard. HealthSnap and the remote dashboard are already in use for remote monitoring at Rush for other programs.

Patients will then start daily blood pressures at home which will automatically be transmitted via the cuff's cellular capabilities to the HealthSnap dashboard. They will continue to have weekly CHW virtual visits during the first month of the program that cover education around blood pressure monitoring compliance, medication adherence, social needs and lifestyle modifications via diet and activity for improvement of CVD risk as per the Heart2Heart Manual created by the Heart2Heart study at Rush. Additionally, directly after enrollment, the patient will receive a virtual visit from the program's nurse (RN) in 48 hours to complete a medication reconciliation. The RN will proceed by remotely monitoring the patient blood pressure readings in the HealthSnap portal. Settings have been created to trigger RN notification for action. These settings include a blood pressure greater than 180/110. In this case, the RN will call the patient and triage the patient for symptoms using the standard of care RN triage model in use in Rush's primary care clinics. If necessary, patient's will be scheduled for clinic follow-up or ED follow-up. Patient's who continue to have stage II hypertension without improvement over 14 days but do not tigger the alerts with elevated pressure, will be monitored at least once every 14 days by the RN, and if not improving, will be forwarded to a remote virtual study pharmacist visit for medication titration.

The study will proceed for a total of 12 weeks, with remote blood pressures recorded for patients daily in the HealthSnap portal. Study goals include improvement of blood pressure to below 130/90 and/or a decrease in systolic blood pressure by 10 mmHg points. If patients reach the goal prior to the end of the study, they will continue with the study until the the completion of the 12-week period, after which they will return to usual care. Patients who do not achieve the goal at the end of the 12-week period will return back to the standard of care model in the primary care clinic. Patients will receive a repeat SDOH screening questionnaire at completion of the study at 12 weeks and on follow-up at a 3-6 month window. A repeat blood pressure will be collected remotely at a 3-6 month window follow-up to assess adherence.

Study goals include enrollment of 150 patients during each 12-week intervention with rolling enrollment. The study will conclude after a 3 year period.

Each of the E3 team members (the CHW, RN, pharmacist, and SW) will document their interactions with the patient in Epic and REDCap as outreach encounters. The encounters will be structured so that important information, such as SDOH screening, race, ethnicity, sex, marital status, zip code, co-morbidities (obesity, diabetes, chronic kidney disease, heart failure, obstructive sleep apnea, and smoking), number of medications, insurer, and number of visits can be data-mined from the Epic notes for analysis. Patient information will be stored in a data base managed by the study data manager and analyst with de-identified patient information.

Data will be analyzed in a pre-intervention and post-intervention manner. Change in blood pressure will be noted, with special attention paid to corresponding changes in SDOH needs based on screening, number of intervention outreaches, and time spent during outreaches. The converse, a lack of a change in blood pressure will also be compared to SDOH needs documented in CHW and social work intervention outreaches as well as successful intervention outreaches.

ELIGIBILITY:
Inclusion Criteria:

* African American and/or Latinx self-identifying
* Stage II hypertension (140/90) or greater
* Following with Rush primary care provider in eligible Rush primary care clinic
* Access to phone or device with video capabilities in the home

Exclusion Criteria:

* Dialysis patient
* Organ transplant recipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Percentage of total participants with improvement of hypertension to below 130/80 mmHg and/or a decrease of 10mmHg in systolic readings | Baseline, 12 weeks
  Percentage of total participants with improvement from stage II hypertension (140/90 mmHg or above) to blood pressure below 130/80 mmHg with home cuff through self monitoring
Percentage of total participants with sustained improvement of blood pressure below 130/80 mmHg at 3-6 month follow-up | 3-6 month follow-up after the 12 week intervention
  Percentage of total participants with sustained improvement of blood pressure below 130/80 mmHg after the intervention at 3-6 month clinic follow-up as measured with a clinic measured blood pressure

SECONDARY OUTCOMES:
Correlation of change in SDOH survey score in relation to hypertension control below 130/80 mmHg | Baseline, 12 weeks
  Does change in survey scores (as measured by decreased total positive points) for pre and post social determinants of health correlate with hypertension control below 130/80 mmHg
Correlation of initial SDOH survey score in relation to hypertension control below 130/80 mmHg | Baseline, 12 weeks
  Does the initial pre intervention survey score for social determinants of health correlate with hypertension control below 130/80 after the intervention at 12 weeks
Correlation of frequency of self monitoring with post intervention ARMS survey scores | Baseline, 12 weeks
  Do higher rates of self monitoring of blood pressure (number of individual blood pressure readings per week) correlate with scores on post intervention ARMS self adherence medication survey scores

CONTACTS AND LOCATIONS:
Overall Officials: David A Ansell, MD, MPH, Principal Investigator — Rush University Medical Center; Laura J Zimmermann, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT06027905/ICF_000.pdf